CLINICAL TRIAL: NCT01015794
Title: Activation of Cervical and Upper Thoracic Brown Adipose Tissue in Humans Via Beta-adrenergic Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 404/09
Record Dates: First submitted 2009-10-29; First posted 2009-11-18 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2009-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Ephedrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adrenergic agonist (Experimental)
  Interventions: Drug: ephedrine hydrochloride

INTERVENTIONS:
Drug: ephedrine hydrochloride — single oral dose, 1mg/kg body weight
Drug: ephedrine hydrochloride — single dose of 1 mg/kg body weight

SUMMARY:
In this study the investigators aim to quantitate the extent of cervical and upper thoracic brown adipose tissue (BAT) activation in lean and obese humans via positron emission tomography-computed tomography (PET-CT) in response to the non-specific beta adrenergic receptor (AR) agonist ephedrine. The investigators hypothesise that this pharmacological adrenergic stimulus will result in activation of BAT in these participants, and that this activation will be reduced in obese patients. This study will provide important preliminary information with respect to allowing the investigators to progress with longer trials with specific beta 3 AR agonists.

ELIGIBILITY:
Inclusion Criteria: healthy group

* Males aged 20 - 40 years
* Free of overt coronary disease (on history, medical examination and ECG)
* Fasting plasma glucose < 6.1 mmol/L and 2 hour OGTT glucose < 7.8 mmol/L
* Unmedicated
* No major illness
* BMI 18 - 25

Inclusion Criteria: obese group

* Males aged 20 - 40 years
* Free of overt coronary disease (on history, medical examination and ECG)
* Unmedicated
* No major illness
* BMI 30+
* Weight < 100 kg
* Height < 185 cm

The inclusion criteria (Obese participants) of body weight less than ~100 kg is implemented as the PET-CT scanner to be utilised (protocol described subsequently) has a limited patient volume. Therefore to fit within the criteria of BMI > 30, only patients of height ~183 cm or less can be recruited, and inclusion of borderline participants will be discussed with co-investigators from the Alfred Hospital Nuclear Medicine Department.

Exclusion Criteria: healthy group

* Unable to give informed consent
* Smokers
* Lactose intolerance

Exclusion Criteria: obese group

* Unable to give informed consent
* Smokers
* Lactose intolerance
* Participant in research projects involving ionising radiation within the past 5 years
* claustrophobia

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2009-12; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
BAT activity via PET-CT | Baseline and 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Alfred Hospital Heart Centre, Prahran, Victoria, Australia

REFERENCES:
- [Result] Carey AL, Formosa MF, Van Every B, Bertovic D, Eikelis N, Lambert GW, Kalff V, Duffy SJ, Cherk MH, Kingwell BA. Ephedrine activates brown adipose tissue in lean but not obese humans. Diabetologia. 2013 Jan;56(1):147-55. doi: 10.1007/s00125-012-2748-1. Epub 2012 Oct 13. PMID 23064293